CLINICAL TRIAL: NCT03195036
Title: Evaluation of an Early Childhood Development Intervention for HIV-Exposed Children in Cameroon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Catholic Relief Services (Other)
Responsible Party: Principal Investigator, Joy Noel Baumgartner, Assistant Research Professor; Director, Evidence Lab, Duke University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D0989; 2017/02/867/CE/CNERSH/SP (Other: Comite National d'Ethique de la Recherche pour la Sante Hum.)
Record Dates: First submitted 2017-06-16; First posted 2017-06-22 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Early Childhood Development in HIV-Exposed Children
Keywords: HIV-exposed; Early Childhood Development; Cameroon

STUDY DESIGN:
Intervention Model Description: This study utilizes a cluster-randomized trial (CRT) design in order to evaluate the impact of the KIDSS ECD program delivered by Catholic Relief Services, specifically the home visiting component, on child development outcomes and utilization of HIV testing services. The main reason for including randomization is to reduce the risk of selection bias. The unit of inference for this CRT is at the individual level but the unit of randomization is the health facility (cluster) level due to issues of program feasibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group of women/children dyads who consent and are patients at the control clinics will not have any exposure to ECD programming.
- Intervention Arm (Experimental): The intervention group of women/children dyads who consent and are patients at the intervention clinics will receive regular home-based ECD services focused on positive parenting and early stimulation.
  Interventions: Behavioral: Home-based ECD services

INTERVENTIONS:
Behavioral: Home-based ECD services — Health facilities will be randomized to intervention and control groups. The clients at clinics assigned to the intervention group will receive Home-based Early Childhood Development (ECD+) program. The clients at clinics assigned to the control group will not receive the Early Childhood Development (ECD) program.
  Other Names: KIDSS Project Home-Based Visits
  Arms: Intervention Arm

SUMMARY:
There is substantial evidence that early childhood development (ECD) programming can improve child health and development outcomes. An important component of ECD programming is supporting positive parenting and early stimulation practices. While many parents could benefit from such programming, mothers that are HIV-infected may particularly benefit given the higher risks of poorer child development among HIV-exposed children. Catholic Relief Services (CRS) in Cameroon is implementing the Key Interventions to Develop Systems and Services (KIDSS) ECD program for HIV-exposed children. This impact evaluation will ascertain to what extent the KIDSS home-based component of the ECD model affects attainment of age-appropriate developmental milestones (measured by the Ages and Stages Questionnaire 3 (ASQ-3)) in HIV-exposed children in Cameroon. The study design is a cluster-randomized controlled trial with a cohort of 200 mother/child dyads across 10 study clinics. HIV+ mothers will be recruited during pregnancy and their children will be followed up until 18 months of age. The intervention group will receive regular home-based ECD services focused on positive parenting and early stimulation. The control group will not have any exposure to ECD services, though they may receive home-based services focused on HIV care and treatment, hygiene, and nutrition. Randomization occurs at the clinic (cluster) level.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Pregnant and currently in 3rd trimester
* Must reside in Nkoldongo district or Djoungolo district
* Willing to be followed up for up to 21 months (pregnancy + postpartum periods)
* Agrees to voluntary participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Attainment of age-appropriate developmental milestones | ASQ-3 score assessed 18 months after birth.
  Child Development Outcomes, measured by ASQ-3 (18-month survey)
Attainment of age-appropriate developmental milestones | ASQ-3 score assessed 12 months after birth.
  Child Development Outcomes, measured by ASQ-3 (12-month survey)
Attainment of age-appropriate developmental milestones | ASQ-3 score assessed 6 months after birth.
  Child Development Outcomes, measured by ASQ-3 (6-month survey)

SECONDARY OUTCOMES:
Attainment of age-appropriate developmental milestones | ASQ-SE score assessed at 18 months after birth.
  Child Development Outcomes, measured by ASQ-Social Emotional (SE)

CONTACTS AND LOCATIONS:
Overall Officials: Joy N Baumgartner, PhD, MSSW, Principal Investigator — Duke University
Locations (1):
- Catholic Relief Services, Yaoundé, Cameroon

IPD SHARING:
Plan to Share IPD: No